Smartphone Addiction Recovery Coach for Young Adults (SARC-YA) Experiment

NCT 1120-0317

December 1, 2020

## [NEW] INFORMED CONSENT TO PARTICIPATE IN RESEARCH (12/1/2020)

Smartphone Addiction Recovery Coach for Young Adults (SARC-YA) Experiment

You are being asked to participate in a study about ways smartphones can support young adults in making positive life choices related to balancing their work or school life with their alcohol or other substance use.

What will happen during the study? You will be randomly placed in 1 of 2 groups. One group will only do interviews. The other group will do interviews and will get a smartphone to use for 6 months. The phones will have surveys and other tools to help with recovery. The surveys will pop up on the phone 5 times a day and ask questions about what you have been doing. They take 2-3 minutes to complete. You will be asked to return the phone at the end of 6 months. Both groups will attend a training focused on ways to support making positive life choices. The group that receives the smartphone will also learn about using the phone and the supportive recovery tools on the phone. All participants will be interviewed at 3, 6, and 9 months postenrollment and may have their urine tested at the interview appointments. Each person will be in the study for 9 months.

What do I have to do if I want to be in the study? To be in the study, you will sign this consent form. The research team will ask you for information that they can use to stay in touch with you. You may be photographed once by project staff or asked to supply one photograph of yourself, and the photograph will be attached to your Locator Form. The photograph will help project staff verify that the person they are interviewing each time is in fact you and not someone else. This photograph is also used to identify and locate you for follow-up interview purposes, and it may be shown to individuals to help locate you. These individuals will only be told that the researchers are trying to locate you for a health study in which you have agreed to participate. At the end of the project and after all follow-up interviews have been completed, a member of the project team will destroy the photograph.

What takes place at an interview? We will ask you questions about how you have been doing for about 30 minutes. You can choose not to answer any question. You will receive a \$75 Visa gift card after the initial interview and training, a \$30 Visa gift card after the completion of each follow up interview (3, 6, and 9 months) and \$15 after each of two office visits, which may be done virtually. You can earn a total of \$195 for participating in the study. You can earn another \$15 visa gift card for referring up to 5 other 18 to 25 year olds who live in McLean County and use alcohol or other drugs at least weekly. This could provide another \$75 in total for referrals.

What are the benefits to me? Being in the study may help support you in making positive life choices or support your recovery. Everyone can earn up to \$195 in gift cards for participating in the study and another \$75 for referring other people, or a total of \$265. If you are in the group that gets the smartphone, you will have unlimited phone calls, texting and a data plan for 6 months. Either way, you will also be helping us learn how smartphones can help other people.

How will my information be shared? Your name and other information that identifies you will be taken out of your file before it is used for analysis and will not be made public. Additionally, we have a **Certificate of Confidentiality** from the National Institutes of Health. This means that we cannot be "forced" to give out any information to anyone that tells them that you are in this study. We would share information about you if you tell us you are going to hurt yourself or someone else or we are made aware of child or elder abuse. However, if you are in the group that gets a smartphone, you should know that:

- a) We cannot protect your confidentiality related to texts, emails and other things you send.
- b) Sending sexual pictures of minors or other inappropriate content to minors is against the law. This can lead to, among other things, prosecution, jail time, and being listed on sex offender registries. By taking our phone, you agree to never send such pictures or inappropriate content. Also, if you receive them from someone else, you will delete them right away.
- c) If you use this phone to send such pictures or other inappropriate content, it will be taken away. Your participation in the study will be ended immediately. We may be ethically and legally obligated to report you to authorities.

What risks am I taking? There is a chance that some information about you could be found out. This is not usually a problem. The staff who work on these studies have been trained and are required to follow federal laws that protect your information. Your interview responses will not be given to family members, counselors or other professionals unless you allow them to see it. After interviews are completed, your answers are combined with those of many other individuals so that when a report is written only group data are reported.

What if I want to quit the study? You may take yourself out of the study at any time by giving a written note to the person who is in charge of the study. If applicable, you will still be able to go to your usual treatment or recovery services. Your answers to questions are important.

| recovery services. Four answers to questions | are important. | | |
|---|---|---|---|
| AGREEMENT TO PARTICIPATE IN THIS ST This study has been explained to me, and I has study. I am aware that I may withdraw from this understand that no one can guarantee or assume involvement in this study will be maintained as research may be reviewed on an anonymous in the study will be maintained as the study will be study will be maintained as the study will be | ive had the opportunity to a<br>is study at any time without<br>ure the results. Confidential<br>coording to federal law. Who | affecting the s<br>ity of records re<br>en required by | ervices I can receive. I<br>elated to my<br>law, the records of the |
| I hereby agree / do not agree (che have received a copy of this consent form for research or project, I can contact Dr. Michael I as a research subject I can contact Dr. Ralph protection of Human Participants at (309) 451. Name and Signature to Participate in the St. | my records. I understand th<br>Dennis at (309) 451-7801, o<br>Weisheit, chair of Chestnut<br>-7855. | at if I have que<br>or if I have que | estions concerning this stions about my rights |
| First and Last Name (please print) | Signature | | Date |
| Witness (signature) | | Date | |
| Ineligible Refused (Reason: | ) | | |